CLINICAL TRIAL: NCT05255640
Title: MULTICENTER OBSERVATIONAL STUDY OF THE OUTCOME OF PATIENTS ADMITTED WITH ACUTE LOWER EXTREMITY ISCHEMIA
Brief Title: OUTCOME OF PATIENTS ADMITTED WITH ACUTE LOWER EXTREMITY ISCHEMIA
Acronym: DEVENIR-IAM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21-PP-27
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Acute Ischemia of Lower Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with ischemia of the lower limbs
  Interventions: Procedure: operation of ischemia of the lower limbs

INTERVENTIONS:
Procedure: operation of ischemia of the lower limbs — The intervention technique is left to the judgment of the investigator to treat the ischemia

SUMMARY:
Acute ischemia of the lower limb (AMI) is a life-threatening emergency that threatens the functional prognosis of the limb. Depending on the clinical presentation and the anatomy of the patient, several therapeutic approaches can be considered: open surgery, endovascular surgery, hybrid surgery or amputation if revascularization is not feasible. The data in the current literature do not allow to clearly establish which therapeutic approach is the most adapted to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years, regardless of gender.
* Diagnosis of AMI defined according to the Rutherford classification (2). AMI may involve one or both lower limbs.
* Be able to understand and give free and informed consent (non-opposition) to participate in the study
* To be affiliated to the social security system
* Not to object to participating in the study (collection of non-objection)

Exclusion Criteria:

* Voluntary discharge of the patient: opposition to the use of the data (withdrawal of the non-objection)
* Termination of the study by decision of the sponsor or investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with lower limb ischemia
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
survival | 30 days
survival | 90 days

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Besançon university hospital, Besançon
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Dijon University Hospital, Dijon
  - Lyon University Hospital, Lyon
  - Nancu University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Nice University Hospital, Nice
  - APHP - Hôpital Mondor, Paris
  - APHP- Ambroise Paré, Paris
  - APHP- Hôpital Bichat, Paris
  - APHP- Hôpital Européen Georges Pompidou, Paris
  - Reims University Hospital, Reims
  - Strasbourg University Hospital, Strasbourg

IPD SHARING:
Plan to Share IPD: No